CLINICAL TRIAL: NCT02919787
Title: Nordic Multicentre Un-blinded Phase II Randomized Controlled Trial (RCT) Evaluating the Additional Efficacy of Adding Chemotherapy Prior to Resection of a Pancreatic Head Malignancy to Avoid Early Mortality in Those Ultimately Resected
Brief Title: Nordic Pancreatic Cancer Trial (NorPACT) - 1
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: St. Olavs Hospital (Other); Haukeland University Hospital (Other); University Hospital of North Norway (Other); Sahlgrenska University Hospital (Other); Karolinska University Hospital (Other); University Hospital, Linkoeping (Other); Lund University Hospital (Other); Odense University Hospital (Other); Helsinki University Hospital, Finland (Unknown); Norrlands University Hospital (Other); Helse Stavanger HF (Other Government)
Responsible Party: Principal Investigator, Knut Jørgen Labori, Senior consultant surgeon, Professor of Surgery, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NorPACT-1; 2015-001635-21 (EudraCT Number)
Record Dates: First submitted 2016-09-14; First posted 2016-09-29 (Estimated); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Pancreatic Cancer
Keywords: Neoadjuvant treatment
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Fluorouracil; Oxaliplatin; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | US Export: No

ARMS (2):
- Surgery and then postoperative adjuvant chemotherapy (Active Comparator): Surgery and then postoperative adjuvant chemotherapy
  Interventions: Procedure: Pancreatic surgery; Drug: 5-FU; Drug: Oxaliplatine; Drug: Irinotecan
- Neoadjuvant chemotherapy, surgery, adjuvant chemotherapy (Experimental): Neoadjuvant chemotherapy, surgery, adjuvant chemotherapy
  Interventions: Drug: 5-FU; Drug: Oxaliplatine; Drug: Irinotecan; Procedure: Pancreatic surgery

INTERVENTIONS:
Drug: 5-FU — Neoadjuvant treatment
  Arms: Neoadjuvant chemotherapy, surgery, adjuvant chemotherapy
Drug: Oxaliplatine — Neoadjuvant treatment
  Arms: Neoadjuvant chemotherapy, surgery, adjuvant chemotherapy
Drug: Irinotecan — Neoadjuvant treatment
  Arms: Neoadjuvant chemotherapy, surgery, adjuvant chemotherapy
Procedure: Pancreatic surgery — All patients
Drug: 5-FU — Adjuvant treatment
Drug: Oxaliplatine — Adjuvant treatment
Drug: Irinotecan — Adjuvant treatment

SUMMARY:
This study evaluate the additional effect of adding chemotherapy prior to resection of a pancreatic head malignancy. The patients will be randomized into two groups; surgery first (control group) and neoadjuvant chemotherapy (intervention). Primary endpoint is overall survival after resection

DETAILED DESCRIPTION:
Pancreatic cancer is the fourth leading cause of cancer-related deaths in Europe and the United States. Surgical resection remains the only potentially curative treatment. However, the median survival of patients undergoing pancreatic resection alone is 16-23 months. The administration of adjuvant chemotherapy leads to an improvement in overall survival. Thus, completion of multimodality treatment (MMT) is the ideal goal and standard of care for treatment of pancreatic ductal adenocarcinoma (PDAC).

Currently, the surgery-first (SF) strategy is the most universally accepted approach to resectable PDAC (and is the standard of care in Norway), but the optimal sequence of surgery and chemotherapy remains unclear.

The purpose of this study is to further investigate the additional efficacy of neoadjuvant chemotherapy to the standard treatment for resectable cancer of the pancreatic head (surgery followed by adjuvant chemotherapy).

ELIGIBILITY:
Inclusion Criteria:

* Resectable adenocarcinoma of the pancreatic head
* T1-3, Nx, M0 (UICC 7th version, 2010)
* Cytologic or histologic confirmation of adenocarcinoma
* Age > 18 year and considered fit for major surgery
* Written informed consent
* Considered able to receive the study specific chemotherapy

Exclusion Criteria:

* Co-morbidity precluding pancreaticoduodenectomy
* Chronic neuropathy ≥ grade 2
* WHO performance score > 2 • Granulocyte count < 1500 per cubic millimetre
* Platelet count < 100 000 per cubic millimeter
* Serum creatinine > 1.5 UNL (upper limit normal range)
* Albumin < 2,5 g/dl
* Female patients in child bearing age not using adequate contraception, pregnant or lactating women • Mental or organic disorders which could interfere with informed consent or treatments
* Other malignancy within the past 5 years, except non-melanomatous skin or non-invasive cervical cancer
* Percutaneous tumor biopsy
* Any reason why, in the opinion of the investigator, the patient should not participate
* Pregnancy
* Breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2016-09 (Actual); Primary Completion 2022-12-22 (Actual); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Overall survival 18 month after randomization | 18 month
  Overall survival at 18 months after date of randomization (intention to treat)

SECONDARY OUTCOMES:
Overall mortality at one year following commencement of allocated treatment. | 1 year
  Overall mortality at one year following commencement of allocated treatment (NT or SF) for those who ultimately undergo resection
Disease-free survival | until 5 years after surgery
  Patient will come to regular after surgery for follow-up visits regarding their disease.
Histopathological response | Arm 1: Baseline and Arm 2; 4 weeks after baseline
  The histopathological response of the tumor to the neoadjuvant treatment will be assessed by established scores (R0 resection and (y)pN0 disease)
Complication rate after surgery | 30 and 90 days
  Complication rate after surgery as measured by Dindo-Clavien/ISPGS classification systems
Feasibility of neoadjuvant and adjuvant chemotherapy | Baseline
  The feasibility of neo-adjuvant and adjuvant chemotherapy measured by common Terminology Criteria for Adverse Events, grade 3-5, dose reduction and dose delay
Health related Quality of Life | until 5 years after surgery
  Data of quality of life will be assessed by the questionnaires EORTC QLQ-30
Health economics | until 5 years after surgery
  Data of quality of life will be assessed by the questionnaires EQ-5D

CONTACTS AND LOCATIONS:
Overall Officials: Knut Jorgen Labori, MD PhD, Principal Investigator — Oslo University Hospital
Locations (13):
- Odense University Hospital, Odense, Denmark
- Helsinki University Hospital, Helsinki, Finland
- Norway (5):
  - Oslo University Hospital, Oslo, Oslo County
  - Haukeland University Hospital, Bergen
  - Stavanger University Hospital, Stavanger
  - Tromsø University Hospital, Stavanger
  - St. Olav University Hospital, Trondheim
- Sweden (6):
  - Sahlgrenska University Hospital, Gothenburg
  - Karolinska University Hospital, Huddinge
  - Linköping University Hospital, Linköping
  - Skåne University Hospital, Lund
  - University Hospital of Umeå, Umeå
  - Uppsala University Hospital, Uppsala

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Labori KJ, Bratlie SO, Andersson B, Angelsen JH, Biorserud C, Bjornsson B, Bringeland EA, Elander N, Garresori H, Gronbech JE, Haux J, Hemmingsson O, Liljefors MG, Myklebust TA, Nymo LS, Peltola K, Pfeiffer P, Sallinen V, Sandstrom P, Sparrelid E, Stenvold H, Soreide K, Tingstedt B, Verbeke C, Ohlund D, Klint L, Dueland S, Lassen K; Nordic Pancreatic Cancer Trial-1 study group. Neoadjuvant FOLFIRINOX versus upfront surgery for resectable pancreatic head cancer (NORPACT-1): a multicentre, randomised, phase 2 trial. Lancet Gastroenterol Hepatol. 2024 Mar;9(3):205-217. doi: 10.1016/S2468-1253(23)00405-3. Epub 2024 Jan 15. PMID 38237621
- [Derived] Labori KJ, Lassen K, Hoem D, Gronbech JE, Soreide JA, Mortensen K, Smaaland R, Sorbye H, Verbeke C, Dueland S. Neoadjuvant chemotherapy versus surgery first for resectable pancreatic cancer (Norwegian Pancreatic Cancer Trial - 1 (NorPACT-1)) - study protocol for a national multicentre randomized controlled trial. BMC Surg. 2017 Aug 25;17(1):94. doi: 10.1186/s12893-017-0291-1. PMID 28841916